CLINICAL TRIAL: NCT02577913
Title: European Active Surveillance Study Comparing Regimens of Administration in Combined Hormonal Contraception
Acronym: EURAS-CORA
Status: Terminated | Type: Observational
Why Stopped: MA of product has been withdrawn from the European market due to stability data
Sponsor: Center for Epidemiology and Health Research, Germany (Other)
Collaborators: Gedeon Richter Plc. (Industry)
Responsible Party: Principal Investigator, Klaas Heinemann, MD, PhD, Dr. Klaas Heinemann, MD PhD MBA, Center for Epidemiology and Health Research, Germany
Other Study IDs: ZEG2014_03
Record Dates: First submitted 2015-10-15; First posted 2015-10-16 (Estimated); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Contraception
Keywords: contraception; contraceptive patch; Levonorgestrel; gestodene; safety

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- FC patch low: Women taking FC Patch low, a transdermal patch releasing 60 micrograms gestodene/24 hours + 13 micrograms ethinyl estradiol/24 hours
- LNG-COC: Women taking levonorgestrel-containing COCs: 1) monophasic preparations containing 20 - 30mcg of ethinylestradiol; 2) multiphasic preparations containing up to 40mcg of ethinylestradiol

SUMMARY:
This study compares the risks of short- and long-term use of FC Patch Low with levonorgestrel-containing combined oral contraceptives (COC-LNG) in a study population representative of the actual users of the individual preparations. FC Patch Low is a transdermal contraceptive patch applied once a week for three consecutive weeks followed by a break of one week (21/7). One patch contains 2.1mg gestodene and 0.55mg ethinyl estradiol, which is equivalent of releasing 0.06mg gestodene and 0.013mg ethinyl estradiol per 24 hours.

DETAILED DESCRIPTION:
FC Patch Low is a transdermal contraceptive patch applied once a week for three consecutive weeks followed by a break of one week (21/7). One patch contains 2.1mg gestodene and 0.55mg ethinyl estradiol, which is equivalent of releasing 0.06mg gestodene and 0.013mg ethinyl estradiol per 24 hours. The most relevant adverse clinical outcome that has been linked to the use of COCs is venous thromboembolism (VTE). Data from randomized clinical trials did not show any serious health concerns for FC Patch Low. However, the statistical power to detect rare adverse events is limited in these studies.

EURAS-CORA is a large, prospective, controlled, long-term active surveillance study to investigate the safety of FC Patch Low with regard to the outcomes of interest. This study follows the European Active Surveillance (EURAS) design methodology with some modifications due to country- and product-specific characteristics. The outcomes of interest will be validated via the attending physicians. A multi-faceted follow-up procedure will ensure a low loss to follow-up rate. This study will involve women from Europe who will be followed for up to 2 years. Data analysis will include multivariable techniques such as Cox regression.

The study has been terminated:

On 10th October, 2016 Gedeon Richter Plc initiated a recall of the FC Patch Low based on stability data provided by Bayer AG (licensor). Under certain conditions the stability tests showed out of specification results. Data from in vitro dissolution tests have shown altered dissolution profile for the gestodene component. Furthermore, visually observable quality defect of crystallization due to the progesterone component (gestodene) had been detected. The clinical relevance of the quality issue is currently not proven. Based on the company's safety database, no increase in the frequency of reported adverse events or in the number of unwanted pregnancies were observed in association with the quality issue of the patch. The Pearl Index calculated based on this post-marketing data and taking into account the possible under-reporting (Pearl Index: 0.50) is considerably lower than the Pearl Index based on the data from clinical trials (Pearl Index: 1.19).

The competent authorities were informed about the quality issue and Gedeon Richter Plc took the precautionary measure to stop marketing and commercializing the product. Wholesale partners were asked to recall the affected product batches currently on the market from pharmacies.

Study investigators were officially informed of the recall and study suspension on 17th October, 2016. The suspension of network expansion activities in Spain and France was immediate. Physician recruitment in Italy had not formally commenced at the time of the study suspension. All relevant ethics committees, including the EMA PAS register, were informed of the study suspension by 21st October, 2016. The maximum duration of contraceptive use for current FC Patch Low users is 10th October 2016 + 3months (or 10th January 2017). Therefore, all women currently enrolled in EURAS-CORA were followed up until January 2017.

On 22nd May 2019, ZEG Berlin were officially notified by Gedeon Richter Plc that FC Patch Low had been withdrawn from the European market.

ELIGIBILITY:
There will be no specific medical inclusion/exclusion criteria and no age restrictions

Inclusion Criteria:

* First ever user of a combined hormonal contraceptive "starter"
* User who restarts a combined hormonal contraceptive after at leat a two month break "restarter"
* Women willing to participate in an active surveillance study

Exclusion Criteria:

- Women who do not understand the major aspects of the study

Min Age: 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women using combined hormonal contraceptives
Sampling Method: Non-Probability Sample
Enrollment: 2281 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2019-05-22 (Actual)

PRIMARY OUTCOMES:
Venous thromboembolism | 24 months
  Deep venous thromboembolism

SECONDARY OUTCOMES:
Arterial thromboembolism | 24 months
  Acute myocardial infarction, cerebrovascular accident, other arterial thromboembolism
Application site reactions | 24 months
  Monitoring of potential skin reactions at the site of Lisvy patch administration
Short- and long-term fertility | 24 months
  return to fertility outcomes after stopping patch use
Pregnancy outcomes | 24 months
  unintended pregnancies during contraceptive use

CONTACTS AND LOCATIONS:
Overall Officials: Klaas Heinemann, MD PhD MBA, Principal Investigator — ZEG Berlin
Locations (1):
- Berlin Center for Epidemiology and Health Research, Berlin, Germany